CLINICAL TRIAL: NCT00634556
Title: Dopaminergic Effects on Cortical Function in Tourette's (Levodopa Protocol)
Acronym: TSfMRI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Other
Other Study IDs: 05-0832; R01MH073856-01A1 (NIH)
Record Dates: First submitted 2008-03-05; First posted 2008-03-13 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Tourette Syndrome
Keywords: Tourette Syndrome; fMRI; levodopa; working memory; dopamine
MeSH Terms: conditions — Tourette Syndrome | interventions — Levodopa; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- levodopa solution 2mg/ml for i.v. use (Experimental): levodopa solution in saline, given intravenously, dosed as per "final protocol" in Black et al 2003.
  Interventions: Drug: levodopa solution 2mg/ml for i.v. use
- Placebo (Placebo Comparator): normal saline i.v.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: levodopa solution 2mg/ml for i.v. use — 2mg/mL in normal saline
  Other Names: L-DOPA; L-3,4-dihydroxyphenylalanine
  Arms: levodopa solution 2mg/ml for i.v. use
Drug: placebo — normal saline
  Other Names: NaCl 0.9% in water
  Arms: Placebo

SUMMARY:
Dr. Kevin J. Black at Washington University is conducting a study to learn whether we can use MRI scans to test dopamine function in the brain and to determine whether the brain performs memory tasks differently in Tourette Syndrome (TS). TS is a movement disorder characterized by vocal tics (sounds) and motor tics (movements). We will measure how and where brain activity changes using magnetic resonance imaging (MRI) scans during memory tasks and after taking levodopa. Levodopa is a drug commonly used for the treatment of Parkinson's disease (PD), a very different movement disorder.

DETAILED DESCRIPTION:
Clinical observations suggest that in TS there is abnormal function in the brain's motor system that can be modified by manipulating dopamine. My colleagues and I have hypothesized that nonmotor brain systems may also show dopamine-sensitive functional abnormalities. Recently we tested this hypothesis using functional magnetic resonance imaging (fMRI). A cognitive task involving working memory (WM) produced excessive activation of several brain regions in TS subjects compared to controls, but this excessive activation normalized after administering the dopamine precursor levodopa (Hershey et al, 2004).

We can state the following focused hypotheses and corresponding specific aims:

(1) In TS, normal performance during a working memory (WM) task requires greater activation of specific brain regions (parietal cortex, medial frontal cortex and thalamus) than in control subjects, and this excess fMRI response is reduced (improved) by exogenous levodopa. (2) These fMRI results in TS relate specifically to WM, to TS, and to dopamine receptor activation, rather than to non-WM components of the cognitive task, comorbidity, placebo effects, or other confounds.

Specific Aim 1. Test whether the preliminary fMRI results generalize to a larger and more representative sample of adults with TS.

Specific Aim 2. Clarify the variables that interact to produce the differential fMRI responses to a WM task and levodopa observed in TS subjects vs controls.

2a. Task components. Control for non-WM components of the task and delineate a "dose-response" curve for effects of WM load on fMRI responses.

2b. Clinical variables. Test whether the fMRI results in our preliminary data are associated with TS itself rather than with comorbid conditions, treatment history, demographic variables, or state variables such as current tic severity / tic suppression.

2c. Pharmacology. Test whether the post-levodopa changes in WM-related fMRI signal relate specifically to levodopa plasma concentration (rather than practice effects, placebo effects, or passage of time) and are replicated by a nonselective dopamine receptor agonist or by a dopamine D2/D3/D4 agonist.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55.
* Tic subjects must meet DSM-IV-TR criteria for a chronic tic disorder.
* Controls are matched for age (within 4 years), sex, handedness (right-handed, non-right-handed), and education (within 2 years), and if possible for race and ethnicity

Exclusion Criteria:

* Inability to give competent informed consent.
* Lactation, pregnancy or possibility of pregnancy.
* Contraindication to MRI (pacemaker; nontrivial metallic foreign bodies; significant claustrophobia).
* Contraindication to levodopa or carbidopa (known allergy).
* Significant neurological disease (not counting the tic disorder).
* Current renal, cardiac or hepatic disease that would make study participation less safe.
* Head injury with loss of consciousness for more than 5 minutes or with neurological sequelae.
* Lifetime history of serious lifetime psychopathology or substance abuse. (Specific exclusions are: lifetime diagnosis of mental retardation, autism, psychosis, mania, somatization disorder, panic disorder, social phobia [excludes symptoms present only when treated with a neuroleptic], anorexia nervosa or bulimia, drug or alcohol dependence, antisocial personality disorder, or dementia, or current major depression.)
* Depot neuroleptics in the past 6 months.
* Other antipsychotics within the past 2 weeks.
* Behavioral therapy for Tics of OCD sx in the past 2 weeks.
* For one half of the subjects in each diagnostic group: any brain-active medications within the past 2 weeks. For the remaining subjects: neuroactive medications in the past 2 weeks other than SSRIs, alpha-2 agonists, norepinephrine reuptake inhibitors, or clonazepam.
* Additional exclusions for controls: No history of tic disorder, OCD or ADHD. If under age 25, no first-degree relative with a tic disorder. No exposure to neuroleptics in the past year and none ever for a period exceeding a week.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2006-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
BOLD (blood oxygen-level dependent) fMRI (functional magnetic resonance imaging) response to a working memory task | From about 30 to 120 minutes after infusion begins

SECONDARY OUTCOMES:
serum prolactin concentration | approximately 2 hours after infusion begins

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J Black, MD, Principal Investigator — Washington Universisty School of Medicine
Locations (1):
- Washington Universisty School of Medicine,, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Vital signs IPD are shared at: Siddiqi SH, Creech ML, Black KJ. Orthostatic stability with intravenous levodopa. PeerJ. 2015 Aug 27;3:e1198. doi: 10.7717/peerj.1198. eCollection 2015. PubMed ID: 26336641 There is no plan to share other IPD.

REFERENCES:
- [Background] Hershey T, Black KJ, Hartlein JM, Barch DM, Braver TS, Carl JL, Perlmutter JS. Cognitive-pharmacologic functional magnetic resonance imaging in tourette syndrome: a pilot study. Biol Psychiatry. 2004 May 1;55(9):916-25. doi: 10.1016/j.biopsych.2004.01.003. PMID 15110735
- [Background] Black KJ, Carl JL, Hartlein JM, Warren SL, Hershey T, Perlmutter JS. Rapid intravenous loading of levodopa for human research: clinical results. J Neurosci Methods. 2003 Jul 15;127(1):19-29. doi: 10.1016/s0165-0270(03)00096-7. PMID 12865145
- [Result] Campbell M, Koller J, Shipley E, Creech M, Hershey T, Black K. Dopaminergic modulation of working memory in Tourette's syndrome [abstract]. J Neuropsychiatry Clin Neurosci 20(2):232, 2008. http://neuro.psychiatryonline.org/article.aspx?articleid=103362
- [Result] Black KJ, Campbell MC, Koller JM, Schneider B, Hershey T. Dopaminergic modulation of working-memory-related cortical activity in Tourette syndrome. Annual meeting, Society for Neuroscience, Chicago, 20 Oct 2009. http://www.sfn.org/
- [Result] Siddiqi SH, Creech ML, Black KJ. Orthostatic stability with intravenous levodopa. PeerJ. 2015 Aug 27;3:e1198. doi: 10.7717/peerj.1198. eCollection 2015. PMID 26336641